CLINICAL TRIAL: NCT03648203
Title: Technology Enabled Asthma Management System (TEAMS) Pilot Study
Acronym: TEAMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: University of Rhode Island (Other)
Responsible Party: Principal Investigator, Jennifer Mammen, Clinical Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SON2018-003
Record Dates: First submitted 2018-07-31; First posted 2018-08-27 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Asthma
Keywords: asthma; quality of life; self-care; healthcare utilization
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: This study is using a single arm, single site, pre-post assessment interventional design, with no control group. Because this is a pilot study, all subjects will receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TEAMS (Experimental): Routine asthma care, as provided in the University of Rochester Medical Center Medicine Clinic, will be augmented by three intervention components over a six-month pilot period : (1) Patient subject smartphone asthma monitoring; (2) Nursing telemedicine follow up (virtual home visits); (3) EMR custom programming to guide nursing assessment and management.
  Interventions: Behavioral: Technology Enabled Asthma Management System

INTERVENTIONS:
Behavioral: Technology Enabled Asthma Management System — See description of arm
  Other Names: TEAMS

SUMMARY:
To evaluate feasibility, acceptability, safety, and preliminary efficacy of a novel patient-centered, technology-based intervention to improve asthma care in younger adult smartphone users.

The program, called TEAMS (Technology Enabled Asthma Management System), uses a combination of smartphone symptom monitoring, guideline-based medication protocols, nursing telemedicine home visits, and Electronic Medical Record (EMR) custom programming.

TEAMS is intended to augment primary asthma care as provided at the University of Rochester Medicine Clinic.

DETAILED DESCRIPTION:
Uncontrolled asthma is a tremendous burden to individuals and society. Asthma is one of the most common chronic health conditions globally, affecting more than 8.2% of adults in the U.S. Of adults with asthma in the U.S., 63% have persistent disease, and less than half are well-controlled. Uncontrolled asthma is associated with bothersome symptoms, economic burden, lost work time, and poorer quality of life. Direct and indirect costs are estimated at 56 billion dollars annually, with over 1.8 million ED visits, 439,000 hospitalizations, and 3,400 deaths in 2010 alone. Asthma morbidity and mortality is preventable. Correct use of controller medication and effective self-management alleviates symptoms, prevents exacerbations, and minimizes long-term damage to lungs associated with pulmonary remodeling. For these reasons, the National Heart Lung & Blood Institute (NHLBI) Guidelines recommend that all individuals with persistent asthma should take daily controller medications and receive consistent self-management training.

Currently, less than half of adults with persistent asthma take controller medication, and most do not self-manage their asthma effectively. Patient, provider, and systems-level factors contribute to this pattern. Patients fail to report symptoms, take medications inconsistently, and have insufficient resources (knowledge, time, transportation, money) to manage their disease.Providers in turn may lack familiarity with current best-practice guidelines, follow alternate prescribing practices, or spend insufficient time educating patients. Translation of asthma management knowledge into practice-based solutions is urgently needed. Many asthma interventions have been implemented within investigator-controlled settings. Problematically, few have been evaluated within or translated into the context of real world practice, and thus hold little benefit for the greater patient population. Limited ability to translate interventions from the bench to clinical settings suggests a need to develop and test interventions within the context in which they are intended to function. Effective real-world intervention to improve asthma outcomes requires development of a multifaceted program targeting key factors at the patient, provider, and systems level.

These include:

* Patient tendency to ignore, forget, and not report symptoms;
* Patient non-adherence to prescribed medication;
* Patient lack of self-management skills and knowledge on how to self-manage effectively;
* Barriers to consistent follow-up (access to care, burdens of time and transportation);
* Provider non-adherence to National Guidelines for step-wise management of asthma; and
* Provider underestimation of symptoms, and lack of time to provide thorough asthma education.

Therefore, the purpose of this study is to test feasibility, acceptability, safety, and preliminary efficacy of comprehensive Technology Enabled Asthma Management System (TEAMS), which addresses these critical factors, in order to improve asthma management and outcomes in younger adults.

The specific aims of the study are:

Aim 1: To evaluate feasibility and acceptability of TEAMS. • Hypothesis A: TEAMS will be feasible for and acceptable to young adults and primary care providers for routine management of asthma, as measured by USE-Q survey data, frequency of symptom self-monitoring and at completion of least one virtual visit, and post-intervention qualitative interviews.

Aim 2: To evaluate safety and preliminary efficacy of TEAMS.

• Hypothesis B: TEAMS will be associated with improved asthma outcomes following intervention, as measured by primary outcomes of: (a) increased asthma control, pulmonary function, quality of life, and secondary outcomes of (b) decreased office visits for asthma exacerbations, asthma-related ED visits, and hospitalizations.

Aim 3: To optimize TEAMS intervention components based on quantitative survey data and qualitative interviews, including patient subject and clinic staff perspectives.

2. STUDY DESIGN

2.1. Overview TEAMS is a multi-level, theoretically-based intervention that capitalizes on patient-provider-nurse partnerships and use of technology to improve the quality and convenience of routine asthma care. TEAMS has Social Cognitive Theory underpinnings. It targets person level factors associated with asthma outcomes (individual knowledge, norms, attitudes, illness beliefs and self-efficacy), self-management behaviors (prevention, monitoring, management and communication of symptoms), and environmental factors (access to care, delivery of guideline-based care).

The overarching goal of TEAMS is to improve asthma outcomes by leveraging capabilities of existing technology (smartphone, telemedicine, electronic medical record). TEAMS will operate in conjunction with standard care in the Medicine Clinic.

ELIGIBILITY:
Inclusion Criteria:

Patient Subjects:

* Target population, Age 18-40; Age criteria may be expanded to include adults older than 40 as needed to meet recruitment needs
* With a diagnosis of intermittent or persistent asthma;
* Possessing an active smartphone with data plan or WiFi access;
* Able to communicate in English.
* Able to perform study-related functions
* Able to give informed consent.

(All patient subjects will be counseled that telemedicine visits consume large amounts of data, and that use of Wifi is recommended. Patient subjects will be required to initial acknowledgement of this in the consent form. Currently however, many people have unlimited data plans, which may allow visits away from Wifi.)

Provider Subjects:

• Primary care provider to patient subjects enrolled in the study

Other Staff Subjects:

• Secretarial or Nursing staff at the clinic, having interaction with patient subjects or procedures.

Exclusion Criteria:

Patient Subjects:

* Diagnosis of confounding respiratory or cardiac diseases (e.g. cystic fibrosis, sarcoidosis, COPD, CHF, Hypertension);
* Pregnancy

Provider Subjects:

• None

Other Staff Subjects:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Acceptability of the TEAMS program for routine asthma management for patients as assessed by USE-Q at end of study | 6 months
  The USE-Q (Usability Satisfaction and Ease of Use Questionnaire) is a 7 point Likert type scale that consists of 21 positive statements which the user rates on a 7-point Likert scale, with 0= strongly disagree to 7=strongly agree.
Change in asthma control from baseline to end of study at 6 months | 6 months
  Clinician-rated asthma control will be measured using the Asthma Control Questionnaire (ACQ) by Juniper. The instrument has 7 questions, each with a range of 0-6 with lower scores representing better asthma control. Total ACQ score is the average of the 7 individual items. A mean score of 0.75 (or less) on the ACQ has a positive predictive value of 0.85 for controlled asthma. A mean score of 1.5 or higher has a positive predictive value of 0.88 for uncontrolled asthma. Minimum important difference (MID) for the ACQ is a change score of 0.5.
Change in Forced Expiratory Volume over 1 second (FEV1) from baseline to end of study at 6 months | 6 months
  FEV1 will be measured using a digital peak flow meter with FEV1 capacity
Change in Asthma-related Quality of life from baseline to end of study at 6 months | 6 months
  Asthma-related quality of life will be measured using the Asthma Quality of Life Questionnaire (AQLQ(S)) by Juniper. The AQLQ measures physical and emotional impact of disease. There are 32 items with a range of 1-7 each, with higher scores representing better quality of life. (7=no impairment; 4= moderate impairment; 1=maximum impairment). The AQLQ consists of 4 domains. Domain scores are computed by averaging the scores of individual items which range from 7 (no impairment) to 1 (maximal impairment). The total AQLQ is computed by averaging the scores across all domains. MID for change in AQLQ total score is 0.5 total, and 0.5 per domain.

SECONDARY OUTCOMES:
Change in frequency of acute healthcare utilization from baseline to end of study at 6 month | 6 months
  Counts (frequency) of asthma-related acute healthcare visits will be extracted from the electronic medical record (ED visits and hospitalizations related to asthma) and will be compared for the equivalent 6 months prior to intervention and the 6 months of intervention
(Qualitative) Participant experiences with and perceptions of TEAMS program | 6 months
  Assessment of participants experiences with and perceptions of the TEAMS program, as assessed by in-depth semi-structured qualitative interview (1:1).

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Gommel, MS, CIM, CIP, Study Director — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mammen JR, Java JJ, Halterman J, Berliant MN, Crowley A, Frey SM, Reznik M, Feldman JM, Schoonmaker JD, Arcoleo K. Development and preliminary results of an Electronic Medical Record (EMR)-integrated smartphone telemedicine program to deliver asthma care remotely. J Telemed Telecare. 2021 May;27(4):217-230. doi: 10.1177/1357633X19870025. Epub 2019 Aug 22. PMID 31438761